CLINICAL TRIAL: NCT02928848
Title: Baseline Performance Predicts tDCS-mediated Improvements in Language Symptoms in Primary Progressive Aphasia
Brief Title: Transcranial Direct Current Stimulation for Primary Progressive Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 818622
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Primary Progressive Aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): Transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation that modulates the resting excitability of neuronal populations, thereby altering patterns of brain activity in potentially behaviorally relevant ways. The stimulation involves 20 minutes of constant stimulation at 1.5 mA.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham tDCS uses identical stimulation parameters as the active condition, however terminates after 30 seconds in order to mimic the sensation of real tDCS.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation that modulates the resting excitability of neuronal populations, thereby altering patterns of brain activity in potentially behaviorally relevant ways. The stimulation involves 20 minutes of constant stimulation at 1.5 mA.

SUMMARY:
In the present sham-controlled study, the investigators examine whether tDCS could be used to enhance language abilities (e.g., picture naming) in individuals with primary progressive aphasia (PPA) primarily characterized by difficulties with speech production.

DETAILED DESCRIPTION:
Primary Progressive Aphasia (PPA) is a neurodegenerative condition characterized by insidious irreversible loss of language abilities. Prior studies suggest that transcranial direct current stimulation (tDCS) directed toward language areas of the brain may help to ameliorate symptoms of PPA. In the current study, the investigators are examining whether tDCS could be used to enhance language abilities (e.g., picture naming) in individuals with PPA variants primarily characterized by difficulties with speech production (non-fluent and logopenic). Participants are being recruited from the Penn Frontotemporal Dementia Center to receive 10 days of both real and sham tDCS (counter-balanced, full-crossover design; participants are naïve to stimulation condition). A battery of language tests are being administered at baseline, immediately post-tDCS (real and sham), and six weeks and twelve weeks following stimulation. Real tDCS may improve language performance in some individuals with PPA. Specifically, the investigators expect that tDCS will be more effective in people whose baseline performance is worse based on previous research. Severity of deficits at baseline may be an important factor in predicting which patients will respond positively to language-targeted tDCS therapies.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 45-80
* Native English speaker
* Diagnosed with Primary Progressive Aphasia
* Subject understands nature of study and able to give informed consent

Exclusion Criteria:

* Cognitive impairment of sufficient severity to preclude giving informed consent
* History of seizures or unexplained loss of consciousness
* Previous craniotomy or any breach of the skull
* Metallic objects in the head or face other than dental braces, fillings or implants
* Pacemaker or implantable cardioverter-defibrillator
* Pregnant

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H B Coslett, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] McConathey EM, White NC, Gervits F, Ash S, Coslett HB, Grossman M, Hamilton RH. Baseline Performance Predicts tDCS-Mediated Improvements in Language Symptoms in Primary Progressive Aphasia. Front Hum Neurosci. 2017 Jun 30;11:347. doi: 10.3389/fnhum.2017.00347. eCollection 2017. PMID 28713256
- See also: Lab website — http://www.med.upenn.edu/lcns/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 10/2017-11/2019. Patients with Primary Progressive Aphasia will be recruited from the clinical practices of Drs. H. Branch Coslett, Roy Hamilton, and Murray Grossman at the Hospital of the University of Pennsylvania. Additional recruitment measures involve flyers posted around the University of Pennsylvania campus and the Hospital of the University of Pennsylvania grounds, as well as online FTD/PPA support groups and in-person support groups around the Philadelphia area.
Pre-assignment Details: 16 participants were enrolled in the study. Subjects were enrolled if they were native English speakers, right handed, and received a diagnosis of primary progressive aphasia (PPA). Note that one participant was diagnosed as having PPA at the time of enrollment; however, it was later learned that this was a misdiagnosis and their data were not analyzed. Baseline Characteristics reported for N=13. The washout period between treatment arms was 12 weeks.
Groups:
- Active tDCS, Then Sham tDCS: Transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation that modulates the resting excitability of neuronal populations, thereby altering patterns of brain activity in potentially behaviorally relevant ways. The active stimulation involves 20 minutes of constant stimulation at 1.5 mA intensity. Following a washout period of 12 weeks after active tDCS in Arm 1, subjects then crossed over to treatment Arm 2, and received sham tDCS.
- Sham tDCS, Then Active tDCS: Sham tDCS uses identical stimulation parameters as the active condition, however terminates after 30 seconds in order to mimic the sensation of active tDCS. Following a washout period of 12 weeks after sham tDCS in Arm 1, subjects then crossed over to treatment Arm 2, and received active tDCS.
Period: Arm 1
Arm/Group | Active tDCS, Then Sham tDCS | Sham tDCS, Then Active tDCS
Started | 9 | 7
Completed | 9 | 6
Not Completed | 0 | 1
Period: Arm 2
Arm/Group | Active tDCS, Then Sham tDCS | Sham tDCS, Then Active tDCS
Started | 9 | 6
Completed | 8 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analyses were conducted on 13 of the 16 people enrolled in the study. Two participants were not included in analyses because they did not complete both arms of the study, and one person was excluded because they were misdiagnosed as having primary progressive aphasia.
Groups:
- Active tDCS, Then Sham: Transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation that modulates the resting excitability of neuronal populations, thereby altering patterns of brain activity in potentially behaviorally relevant ways. The active stimulation condition involves 20 minutes of constant stimulation at 1.5 mA. Arm 1 data were collected prior to active tDCS, whereas Arm 2 data reflect performance 12 weeks following active tDCS (prior to crossing over to the sham tDCS treatment arm).
- Sham tDCS, Then Active: Sham tDCS uses identical stimulation parameters as the active condition, however terminates after 30 seconds in order to mimic the sensation of real tDCS. Arm 1 data were collected prior to sham tDCS, whereas Arm 2 data reflect performance 12 weeks following sham tDCS (prior to crossing over to the active tDCS treatment arm).
- Total: Total of all reporting groups
Arm/Group | Active tDCS, Then Sham | Sham tDCS, Then Active | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.29 (7.67) | 66.33 (6.18) | 66.31 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
Western Aphasia Battery - Aphasia Quotient (WAB-AQ) [Mean (Standard Deviation); unit: units on a scale] — The WAB-AQ is a weighted average of all subtest scores relating to spoken language, measuring language ability. It is a sum of all subtest scores from the first part of the WAB (Spontaneous speech, Auditory verbal comprehension, Repetition, Naming and word finding). We report the total average score and standard deviation. The total range is 0-100 (higher scores indicating better performance).
  units on a scale
    Arm 1 | 79.84 (9.68) | 85.55 (7.80) | 82.38 (9.61)
    Arm 2 | 78.39 (9.24) | 85.55 (7.02) | 81.23 (10.10)

OUTCOME MEASURES:

1. Primary Outcome: Aphasia Severity (WAB-AQ): Effects of Active tDCS (Baseline vs. 0 Weeks Immediately Following Stimulation)
Description: The Western Aphasia Battery (WAB) was administered at baseline and immediately post-tDCS (real; sham) following the termination of the tDCS session on the same day (0 week). We computed WAB-Aphasia Quotient (WAB-AQ), a measure of overall aphasia severity with higher scores indicating better language performance. The WAB assesses the following language domains in subtests: fluency, comprehension, repetition, and naming. We examined change in WAB-AQ and each of the sub-tests from baseline. Difference scores were computed by subtracting the post-intervention score (0 weeks) from baseline for each study arm to assess the impact of real/active vs sham tDCS on severity and each sub-test. Scale title: WAB-AQ; scale values: 0-100; higher scores=better outcome.
Time Frame: Difference in WAB-AQ from Baseline at 0-weeks Post-stimulation
Population: Participants who completed both arms of the study to the 0-week follow-up (N=13). Of the 16 participants enrolled, 3 were excluded from the 0-week follow-up for the following reasons: withdrew prior to starting treatment arm 1 (n=2) and misdiagnosed as PPA (n=1).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS, Then Sham tDCS | Sham tDCS, Then Active tDCS
Number analyzed (Participants) | 7 | 6
score on a scale
  Arm 1: 0 Week Follow-up | 2.68 (2.04) | .87 (2.83)
  Arm 2: 0 Week Follow-up | 1.98 (2.75) | 2.25 (2.04)
Statistical Analysis 1: Comparison: Active tDCS, Then Sham tDCS vs Sham tDCS, Then Active tDCS; Repeated-measures analysis of variance (RM-ANOVA) with Condition (active, sham) and time point (baseline, 0-week) as within-subject factors. Analysis tests whether active vs. sham stimulation confers a greater improvement in overall language ability, as measured by the Western Aphasia Battery Aphasia Quotient (WAB-AQ), that endures over time; Test type: Other; p = 0.14, ANOVA — The a priori threshold for statistical significance was p < .05

2. Secondary Outcome: Naming Ability (WAB Naming Subtest): Effects of Active tDCS Baseline vs. 0 Weeks Immediately Following Stimulation
Description: WAB-naming subtest used common objects as stimuli. Participants were required to name the objects. Three-point maximum score could be earned for each stimulus and a total of 60-points could be earned on this task; points were deducted if the response was incorrect and required a cue or if the response included a paraphasia.
Time Frame: Difference in WAB Naming Subtest from Baseline at 0-weeks Post-stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active tDCS, Then Sham tDCS: Transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation that modulates the resting excitability of neuronal populations, thereby altering patterns of brain activity in potentially behaviorally relevant ways. The active stimulation involves 20 minutes of constant stimulation at 1.5 mA intensity.
- Sham tDCS, Then Active tDCS: Sham tDCS uses identical stimulation parameters as the active condition, however terminates after 30 seconds in order to mimic the sensation of active tDCS.
Arm/Group | Active tDCS, Then Sham tDCS | Sham tDCS, Then Active tDCS
Number analyzed (Participants) | 7 | 6
score on a scale
  Arm 1: 0-week Follow-up | .63 (.49) | .11 (.59)
  Arm 2: 0-week Follow-up | .26 (.83) | .63 (.35)
Statistical Analysis 1: Comparison: Active tDCS, Then Sham tDCS vs Sham tDCS, Then Active tDCS; Repeated-measures analysis of variance (RM-ANOVA) with Condition (active, sham) and time point (baseline, 0-weeks) as within-subject factors. Analysis tests whether active vs. sham stimulation confers a greater improvement in naming ability, as measured by the naming subtest of the WAB, that endures over time; Test type: Other; p = .02, ANOVA — The a priori threshold for statistical significance was p < .05

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events are reported to the PI and IRB within 24-48 hours of the initial event.
Groups:
- Active tDCS: Transcranial direct current stimulation (tDCS) is a type of noninvasive brain stimulation that modulates the resting excitability of neuronal populations, thereby altering patterns of brain activity in potentially behaviorally relevant ways. The active stimulation involves 20 minutes of constant stimulation at 1.5 mA intensity.
- Sham tDCS: Sham tDCS uses identical stimulation parameters as the active condition, however terminates after 30 seconds in order to mimic the sensation of active tDCS.
Arm/Group | Active tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Withdrawal of two participants resulted in 14/16 who completed at least one treatment arm; additional participants were excluded due to not completing both treatment arms (N=2) and misdiagnosis (N=1). Data analyzed for N=13 participants for baseline to 0-week post-stimulation. One participant's second treatment arm was delayed by one week.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT02928848/Prot_SAP_000.pdf